CLINICAL TRIAL: NCT01266473
Title: Efficacy Study of Physiotherapy for Airway Clearance in Cystic Fibrosis. Randomized Controlled Trials in Single Subjects (N of 1 RCT's).
Brief Title: Study of Individualized Physiotherapy for Airway Clearance in Cystic Fibrosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010/802
Record Dates: First submitted 2010-09-06; First posted 2010-12-24 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Cystic Fibrosis
Keywords: Adults
MeSH Terms: conditions — Cystic Fibrosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physiotherapy techniques (Experimental): Cough Technique vs Forced Expiration Technique
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy for Airway Clearance

SUMMARY:
The purpose of this study is to investigate individual efficacy in Physiotherapy for Airway Clearance, and to investigate user experience, i.e.utility value and preference.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: CF
* Age >18 years
* Amount of sputum >5 ml/60 min
* Wet inhalation of saline/DNase/both
* Informed consent

Exclusion Criteria:

* Respiratory failure
* Hemoptysis
* Bacteriology (burkholderia cephacia, multi-resistent pseudomonas aeruginosa, atypical mycobacteria, MRSA).
* Ongoing intravenous medication
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Expectorated sputum (gram) | 8 weeks
  Total amount of expectorated sputum (g) will be collected and weighed wet after each intervention for eight weeks, using a Mettler TOLEDO Weighing Balance (EL 202, accuracy: 0.01 g).
  N of 1 trial design. Each trial consist of eight pairs (8 weeks) of treatment periods with two interventions each week (one with Cough Technique and one with Forced Expiration technique), 16 treatments for each participant. Outcome measure after each treatment.

SECONDARY OUTCOMES:
Patient's experience, i.e. perceived utility value and preference of technique. | 8 weeks
  Utility value: Measured by self-reported questionnaire after completion of each intervention in week 8.
  Preference: Measured by three self-reported questions after both interventions in week 8.

OTHER OUTCOMES:
Physiological measurements | 8 weeks
  Oxygen saturation and heart rate measurements in the beginning and at the end of each intervention.
  Pulmonary function tests (week 2): measurements before and after each intervention with spirometry.
Health related quality of life (HRQOL) | 8 weeks
  HRQOL measured by the Cystic Fibrosis Questionnaire Revised (CFQR-R), i.e. respiratory symptoms, in the beginning and at completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Gursli, PT, MSc, Principal Investigator — Oslo University Hospital, National Centre for cystic fibrosis

REFERENCES:
- [Derived] Gursli S, Quittner A, Jahnsen RB, Skrede B, Stuge B, Bakkeheim E. Airway clearance physiotherapy and health-related quality of life in cystic fibrosis. PLoS One. 2022 Oct 18;17(10):e0276310. doi: 10.1371/journal.pone.0276310. eCollection 2022. PMID 36256673